CLINICAL TRIAL: NCT00446147
Title: Double-Blind Phase III Study of Pyridoxine vs Placebo for the Prevention of Capecitabine-induced Hand-Foot Syndrome
Brief Title: Study of Pyridoxine for Hand-Foot Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Oncologist, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AMC-ONCGI-0403
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Results first posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-01

CONDITIONS: Hand-foot Syndrome
Keywords: hand-foot syndrome; capecitabine; pyridoxine; prevention
MeSH Terms: conditions — Hand-Foot Syndrome | interventions — Pyridoxine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): one tablet twice per day, which is identical to pyridoxine
  Interventions: Drug: Placebo
- Pyridoxine (Experimental): 100 mg twice per day
  Interventions: Drug: Pyridoxine

INTERVENTIONS:
Drug: Pyridoxine — 100mg BID/daily, Per oral
  Arms: Pyridoxine
Drug: Placebo — placebo 100mg BID/daily, Per oral
  Arms: Placebo

SUMMARY:
Although pyridoxine has been used empirically for the prevention of capecitabine associated hand-foot syndrome (HFS), its efficacy needs to be demonstrated in prospective controlled trials. The investigators therefore performed a prospective randomized double-blind study to determine whether pyridoxine 200 mg/day can prevent the development of HFS when given concurrently with capecitabine. The investigators also tested the ability of pyridoxine to treat primary occurrence of grade 2-3 HFS.

DETAILED DESCRIPTION:
Although pyridoxine has been used empirically for the prevention of capecitabine associated HFS, its efficacy needs to be demonstrated in prospective controlled trials. We estimated that the HFS rate with placebo and pyridoxine would be 0.35 and 0.18, respectively, and we therefore calculated that a sample size of 345 patients would be necessary to detect these hazard rates with an 80% power (β=0.2) and two-sided significance level of α=0.05. We assumed a follow up loss rate of 10%, thus requiring 380 patients to be randomized. Chemotherapy-naive patients with gastrointestinal tract cancers who were scheduled for capecitabine-containing chemotherapy were assigned to receive oral pyridoxine or placebo in randomized double-blind placebo controlled study. Pyridoxine 100 mg b.i.d was prescribed to the patients in the pyridoxine group, identical placebo 100 mg b.i.d was prescribed in the placebo group by the closed envelop randomization. Patients were stratified by chemotherapy regimen: capecitabine alone (X), capecitabine and cisplatin (XP), or docetaxel, capecitabine, and cisplatin (DXP). Patients were observed until NCI CTC grade 2 or 3 HFS developed or capecitabine-containing chemotherapy ended. Patients in the placebo group who developed grade 2 or 3 HFS were randomized to receive pyridoxine or placebo for the next chemotherapy cycle to determine whether pyridoxine could improve HFS, and the same treatment was continued for 2 chemotherapy cycles.

ELIGIBILITY:
Inclusion Criteria:

* Gastrointestinal tract cancer patients treated with capecitabine-containing chemotherapy as a first-line treatment were randomly allocated to concurrent treatment with pyridoxine or placebo.
* All patients were 18 to 70 years old
* Had Eastern Cooperative Oncology Group (ECOG) performance status of 2 or lower
* An estimated life expectancy > 3 months
* Adequate bone marrow function, including white blood cell (WBC) count of >3500 cells/㎕ and platelet count of >100000/㎕
* Adequate renal function (serum creatinine concentration <1.5 mg/㎗)
* Adequate liver function with (serum bilirubin concentration <1.5 mg/㎗, transaminase <3 times the upper normal limit, and serum albumin >2.5 mg/㎗).

Exclusion Criteria:

* Previous treatment for HFS
* Hypersensitivity to pyridoxine
* A combination of other malignancies
* Serious illnesses or medical conditions
* Immune suppression or positive human immunodeficiency virus (HIV) serology
* Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2004-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, Principal Investigator — Asan Medical Center IRB

REFERENCES:
- [Derived] Kang YK, Lee SS, Yoon DH, Lee SY, Chun YJ, Kim MS, Ryu MH, Chang HM, Lee JL, Kim TW. Pyridoxine is not effective to prevent hand-foot syndrome associated with capecitabine therapy: results of a randomized, double-blind, placebo-controlled study. J Clin Oncol. 2010 Aug 20;28(24):3824-9. doi: 10.1200/JCO.2010.29.1807. Epub 2010 Jul 12. PMID 20625131

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Pyridoxine
Started | 195 | 194
Completed | 180 | 180
Not Completed | 15 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pyridoxine | Total
Number analyzed (Participants) | 180 | 180 | 360
Age, Customized [Median (Full Range); unit: years]
  Age_median | 56 [28 to 74] | 56 [20 to 75] | 56 [20 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 59 | 135
  Male | 104 | 121 | 225
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 180 | 180 | 360

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Dose of Capecitabine Until the Development of Grade 2 or Higher Hand-foot Syndrome
Description: A total administered dose of capecitabine until the development of grade 2 or higher hand-foot syndrome during the chemotherapy.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: miligram per square meter
Arm/Group | Placebo | Pyridoxine
Number analyzed (Participants) | 180 | 180
miligram per square meter | 70000 [69384 to 70615] | 70000 [60010 to 79989]

2. Secondary Outcome: Number of Patients With Hand-foot Syndrome
Description: Number of patients with any grade of hand-foot syndrome
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Placebo | Pyridoxine
Number analyzed (Participants) | 180 | 180
participants | 55 | 57

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Placebo | Pyridoxine
Serious Adverse Events (participants affected / at risk) | 0/180 | 0/180
Other Adverse Events (participants affected / at risk) | 0/180 | 0/180

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No